CLINICAL TRIAL: NCT02895230
Title: Androgen-Deprivation Therapy and Cardiovascular Risk: A Nationwide Population-based Cohort Study
Acronym: ADTCR
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC13_8812
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer; Androgen-deprivation Therapy
Keywords: Androgen-deprivation therapy; Prostate cancer; Nationwide population-based cohort; Myocardial infarction; Ischemic stroke
MeSH Terms: conditions — Prostatic Neoplasms; Myocardial Infarction; Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Men with prostate cancer with androgen-deprivation therapy: Using the French Health Reimbursement Agency database and French hospital discharge database, the investigators will identify all men with prostate cancer who had either, at least one dispensation in a 1.5-year period (1st July 2010 to 31st December 2011) of an androgen-deprivation therapy or a hospitalization for orchiectomy. The French Health Insurance System covers the entire French population (65.3 million inhabitants in 2012).
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — An extraction from French Health Reimbursement Agency database and French hospital discharge database will be performed using a simplified request based on inclusion criteria but the extraction will encompass a 4-year period to ensure sufficient follow-up.

SUMMARY:
The research focuses on the safety profile of androgen-deprivation therapy (ADT). The hypothesis is that safety issue, as regards to cardiovascular risk, is not homogenous across the spectrum of androgen-deprivation therapy modalities. Our study will encompass all ADT modalities including intermittent ADT.

ADT is a cornerstone therapy in prostate cancer management. Decisions about ADT should weigh improvements in cancer-specific outcomes against potential increased risks for cardiovascular diseases. The potential for harm from ADT should be more precisely defined according to the type of ADT. Those potential risks underscore the importance of better understanding benefits of ADT, especially in contexts where data are still lacking.ADT is also indicated in sexually deviant behavior.

DETAILED DESCRIPTION:
Our study is a nationwide population-based prospective cohort on 4 years thanks to the French Health Reimbursement Agency database (Système National d'Information Inter-Régimes de l'Assurance Maladie, SNIIRAM) and French hospital discharge database (Programme de Médicalisation des Systèmes d'Information; PMSI). A unique civil registration number has been assigned to all French residents and this number unambiguously links those two databases.

ELIGIBILITY:
Inclusion Criteria:

* Adults men, age greater 18 years,
* Affiliation to French Health System,
* Diagnosis of prostate cancer
* At least one dispensation (leading to a reimbursement claim) in a 1.5 year period of an androgen-deprivation therapy or a hospitalization for orchiectomy.

Exclusion Criteria:

* Orchiectomy for another reason that prostate cancer.
* Patients treated with both Gonadotropin Releasing Hormone agonists and bilateral orchiectomy will be excluded from analyses.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using the French Health Reimbursement Agency database and French hospital discharge database, the investigators will identify all men with prostate cancer who had either, at least one dispensation in a 1.5-year period of an androgen-deprivation therapy or a hospitalization for orchiectomy. The French Health Insurance System covers the entire French population (65.3 million inhabitants in 2012).
Sampling Method: Non-Probability Sample
Enrollment: 38690 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Association between androgen-deprivation therapy and vascular stroke | 2 years after the beginning of androgen-deprivation therapy
  To investigate the association between different modalities of androgen-deprivation therapy (continuous or intermittent use of Gonadotropin Releasing Hormone (GnRH) agonists, GnRH antagonists, oral antiandrogens, or orchiectomy) and myocardial infarction or ischemic stroke in French men with prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel OGER, MD, PhD, Study Director — CHU Rennes
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scailteux LM, Vincendeau S, Balusson F, Leclercq C, Happe A, Le Nautout B, Polard E, Nowak E, Oger E. Androgen deprivation therapy and cardiovascular risk: No meaningful difference between GnRH antagonist and agonists-a nationwide population-based cohort study based on 2010-2013 French Health Insurance data. Eur J Cancer. 2017 May;77:99-108. doi: 10.1016/j.ejca.2017.03.002. Epub 2017 Apr 5. PMID 28390298
- [Result] Scailteux LM. Response to letter - Androgen deprivation therapy and cardiovascular risk: No meaningful difference between GnRH antagonist and agonists. Eur J Cancer. 2017 Dec;87:204. doi: 10.1016/j.ejca.2017.06.042. Epub 2017 Jul 26. No abstract available. PMID 28756060